CLINICAL TRIAL: NCT03166683
Title: Standard of Care Versus a New Collagen and Polyethylene Glycol Haemostatic/Sealant Patch (Hemopatch) During Liver Resection. A Multicentre, Non-inferiority Prospective Randomized Study (IBERLIVER-study)
Brief Title: Standard of Care Versus Hemopatch® During Liver Resection
Acronym: IBERLIVER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IBERLIVER
Record Dates: First submitted 2017-04-04; First posted 2017-05-25 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-11

CONDITIONS: Liver Cancer; Hemorrhage Liver; Bile Leak; Surgery; Tumor Liver
MeSH Terms: conditions — Liver Neoplasms; Carcinoma, Hepatocellular | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: Prospective, randomized (1:1) study of 2 treatment groups (hemopatch versus standard of care) in liver resection surgery. Non-inferiority study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemopatch (Experimental): Use of hemopatch like a control of bile leakage/sealant during liver resection surgery.
  Interventions: Other: Hemopatch
- Standard of care (Active Comparator): Application of standards of care, may include other sealant / hemostatic devices as patches or liquid/gels, during liver resection surgery.
  Interventions: Other: Standard of care

INTERVENTIONS:
Other: Hemopatch — Liver resection surgery with collagen and polyethylene glycol haemostatic/sealant patch placement
  Arms: Hemopatch
Other: Standard of care — Standard of care include other sealant / hemostatic devices as patches or liquid/gels
  Arms: Standard of care

SUMMARY:
This multicentre prospective and randomized study aims to compare the sealant effect after surgical liver resection of a new collagen - polyethylene glycol hemostatic / sealant patch (Hemopatch) vs standard of care.

DETAILED DESCRIPTION:
Liver resection is the only potentially curative treatment in malignant or benign hepatobiliary lesions. Biliary leakage is a postoperative complication (5-10%) which may have considerable consequences. Surgical techniques and devices to facilitate the control of bile leakage have been developed in the last decades and have minimized operative risks of liver resection. Nevertheless, hepatic parenchymal transection can be associated with bile leakage due to the division of small ducts. In order to achieve control over parenchyma from the section surface and to prevent intraperitoneal complications attributed to bile leakage/bleeding various locally applicable agents are in use. This control of bile leakage include fibrin sealant and synthetic glues. Evidence from randomized controlled trials regarding the use of fibrin sealants on their own or combined with a collagenfleece has shown Little efficacy.

A new collagen and polyethylene glycol hemostatic/sealant patch (Hemopatch) [Baxter, Vienna, Austria] is indicated for local hemostasis of capillary bleeding and bleeding of parenchymal organs. The felt structure being rich in surface gives a framework for the adhesion of blood platelets, thus providing an additional impetus as a sealant agent.

The investigators aim to demonstrate the sealing capability of hemopatch and to prove its non-inferiority to the standard of care (may include other sealant / hemostatic devices as patches or liquid/gels). There will be 2 groups to compare. The study group where Hemopatch is applied at the end of surgery. And the control group, where standard of care measures will be applied at the end of surgery. The end-point is the assessment of control of bile leakage at 1, 2, 3, and 4 day, during the hospital stay and or at 30 days for both treatment group. The secondary end-points are bleeding complications (re-bleeding, hematoma formation), volume of fluid drained on day 1 to day 4 after surgery, hemoglobin variation from pre-operative until discharge and post-operatory complications until 30th day pos-op.

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years.
* Patients with an indication for open liver resection (segmental or non-segmental).
* Target bleeding site of generalized bleeding that persists on the cut surface of the liver in which hemostasis cannot be achieved by conventional methods.
* Willing and able to complete the clinical trial procedures, as described in the protocol.
* Signed written informed consent to participate in this clinical trial.

Exclusion Criteria:

* Presence of coagulation disorder, Klatskin tumour. Cirrhosis, re-hepatectomies and biliary resections
* Concurrent participation in another clinical trial with a medical device or medicinal product or with interfering endpoints.
* Concurrent or previous therapy with systemic pharmacologic agents promoting blood clotting including but not limited to tranexamic acid, activated factor VII, fibrinogen and aprotinin.
* Known allergy or hypersensitivity to a component of the investigational treatments Hemopatch® ,to riboflavin or to proteins of bovine origin.
* Pregnancy or breast-feeding.
* Inability to understand the nature and the extent of the trial and the procedures required.

Criteria to be checked during surgery (intraoperative exclusion criteria):

* Infected wound area.
* Persistent major bleeding after primary hemostasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 284 (Estimated)
Dates: Start 2017-12 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Control of bile leakage | From day 1 to day 4
  analysis of bilirubin (mg/dL),in the drain fluid

SECONDARY OUTCOMES:
Bleeding | From the surgery day until day 30
  Total volume of blood, quantified though aspiration and drainage (Quantification of total number of deciliters (dL) of blood gathered)
Analysis of hemoglobin | From the surgery day until day 30
  Quantification of hemoglobin (mg/dL), in the drain fluid
Bleeding complications | From the surgery day until day 30
  Presence (YES or NO compatible imagen of hemorrhage )of post-hepatectomy hemorrhage or Hematoma formation (Valid imaging tests of presence or absence can be checked by : abdomen ecography, TAC or RNM)
Transfusion requirements | From the surgery day until day 30
  Quantification of number of packed red blood cells

OTHER OUTCOMES:
Bile leakage severity | From the surgery day until day 30
  Classification A,B,C. According to International Study Group of Liver Surgery (ISGLS)
Morbidity | From the surgery day until day 30
  * Postoperative Ileus (refers to obstipation and intolerance of oral intake due to non mechanical factors that disrupt the normal coordinated propulsive motor activity of the gastrointestinal tract following abdominal or non abdominal surgery)
  * Allergic reaction (Signs and symptoms are urticarial rash; pruritus; flushing; angioedema of the face, extremities, or laryngeal tissues (leading to throat tightness with stridor, or rarely asphyxiation); wheezing; gastrointestinal symptoms; and/or hypotension after use Hemopatch)
  * Intrabdominal Infection (It describes a diverse set of diseases. It is broadly defined as peritoneal inflammation in response to microorganisms, resulting in purulence in the peritoneal cavity.)
Mortality | From the surgery day until day 30
  Death: number of patients dying during study

CONTACTS AND LOCATIONS:
Overall Officials: Miguel Angel Gómez Bravo, PhD, Principal Investigator — Hospitales Universitarios Virgen del Rocío

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data for IPD is planned to be shared with all participants within 6 months of data completion
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 12 MONTHS

REFERENCES:
- [Background] Baumgartner B, Draxler W, Lewis KM. Treatment of Severe Aortic Bleeding Using Hemopatch in Swine on Dual Antiplatelet Therapy. J Invest Surg. 2016 Dec;29(6):343-351. doi: 10.3109/08941939.2016.1154627. Epub 2016 Mar 22. PMID 27002742
- [Background] Erdogan D, Busch OR, van Delden OM, Rauws EA, Gouma DJ, van Gulik TM. Incidence and management of bile leakage after partial liver resection. Dig Surg. 2008;25(1):60-6. doi: 10.1159/000118024. Epub 2008 Feb 22. PMID 18292662
- [Background] Figueras J, Llado L, Miro M, Ramos E, Torras J, Fabregat J, Serrano T. Application of fibrin glue sealant after hepatectomy does not seem justified: results of a randomized study in 300 patients. Ann Surg. 2007 Apr;245(4):536-42. doi: 10.1097/01.sla.0000245846.37046.57. PMID 17414601
- [Background] Guillaud A, Pery C, Campillo B, Lourdais A, Sulpice L, Boudjema K. Incidence and predictive factors of clinically relevant bile leakage in the modern era of liver resections. HPB (Oxford). 2013 Mar;15(3):224-9. doi: 10.1111/j.1477-2574.2012.00580.x. Epub 2012 Oct 4. PMID 23374363
- [Background] Lewis KM, McKee J, Schiviz A, Bauer A, Wolfsegger M, Goppelt A. Randomized, controlled comparison of advanced hemostatic pads in hepatic surgical models. ISRN Surg. 2014 Mar 4;2014:930803. doi: 10.1155/2014/930803. eCollection 2014. PMID 24729905
- [Background] Lewis KM, Schiviz A, Hedrich HC, Regenbogen J, Goppelt A. Hemostatic efficacy of a novel, PEG-coated collagen pad in clinically relevant animal models. Int J Surg. 2014;12(9):940-4. doi: 10.1016/j.ijsu.2014.07.017. Epub 2014 Aug 6. PMID 25106082
- [Background] Lewis KM, Spazierer D, Slezak P, Baumgartner B, Regenbogen J, Gulle H. Swelling, sealing, and hemostatic ability of a novel biomaterial: A polyethylene glycol-coated collagen pad. J Biomater Appl. 2014 Nov;29(5):780-8. doi: 10.1177/0885328214545500. Epub 2014 Aug 1. PMID 25085811
- [Background] Rahbari NN, Garden OJ, Padbury R, Maddern G, Koch M, Hugh TJ, Fan ST, Nimura Y, Figueras J, Vauthey JN, Rees M, Adam R, Dematteo RP, Greig P, Usatoff V, Banting S, Nagino M, Capussotti L, Yokoyama Y, Brooke-Smith M, Crawford M, Christophi C, Makuuchi M, Buchler MW, Weitz J. Post-hepatectomy haemorrhage: a definition and grading by the International Study Group of Liver Surgery (ISGLS). HPB (Oxford). 2011 Aug;13(8):528-35. doi: 10.1111/j.1477-2574.2011.00319.x. Epub 2011 Jun 7. PMID 21762295
- [Background] Nagano Y, Togo S, Tanaka K, Masui H, Endo I, Sekido H, Nagahori K, Shimada H. Risk factors and management of bile leakage after hepatic resection. World J Surg. 2003 Jun;27(6):695-8. doi: 10.1007/s00268-003-6907-x. Epub 2003 May 13. PMID 12732991
- [Background] Ruggiero R, Docimo L, Tolone S, De Palma M, Musella M, Pezzolla A, Gubitosi A, Parmeggiani D, Pirozzi R, Gili S, Parisi S, D'Alessandro A, Docimo G. Effectiveness of an advanced hemostatic pad combined with harmonic scalpel in thyroid surgery. A prospective study. Int J Surg. 2016 Apr;28 Suppl 1:S17-21. doi: 10.1016/j.ijsu.2015.12.044. Epub 2015 Dec 17. PMID 26708861
- [Background] Sadamori H, Yagi T, Matsuda H, Shinoura S, Umeda Y, Fujiwara T. Intractable bile leakage after hepatectomy for hepatocellular carcinoma in 359 recent cases. Dig Surg. 2012;29(2):149-56. doi: 10.1159/000337313. Epub 2012 May 3. PMID 22555445
- [Background] Sakamoto K, Tamesa T, Yukio T, Tokuhisa Y, Maeda Y, Oka M. Risk Factors and Managements of Bile Leakage After Hepatectomy. World J Surg. 2016 Jan;40(1):182-9. doi: 10.1007/s00268-015-3156-8. PMID 26159119
- [Background] Tanaka S, Hirohashi K, Tanaka H, Shuto T, Lee SH, Kubo S, Takemura S, Yamamoto T, Uenishi T, Kinoshita H. Incidence and management of bile leakage after hepatic resection for malignant hepatic tumors. J Am Coll Surg. 2002 Oct;195(4):484-9. doi: 10.1016/s1072-7515(02)01288-7. PMID 12375753
- [Background] Weltert L, D'Aleo S, Chirichilli I, Falco M, Turani F, Bellisario A, De Paulis R. Prospective Randomized Clinical Trial of HEMOPATCH Topical Sealant in Cardiac Surgery. Surg Technol Int. 2016 Oct;XXIX:sti29/756. Epub 2016 Jul 29. PMID 27466878
- [Background] Yamashita Y, Hamatsu T, Rikimaru T, Tanaka S, Shirabe K, Shimada M, Sugimachi K. Bile leakage after hepatic resection. Ann Surg. 2001 Jan;233(1):45-50. doi: 10.1097/00000658-200101000-00008. PMID 11141224